CLINICAL TRIAL: NCT06349928
Title: "The Show Must go on". The Experience of Injuries Among Dancers: Fears, Thoughts, and Beliefs. A Qualitative Study
Brief Title: "The Show Must go on" : The Experience of Injuries Among Dancers: Fears, Thoughts, and Beliefs. A Qualitative Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Elisabetta Bigi, Physiotherapist, University of Siena
Other Study IDs: MASF_Dancers01
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Injuries; Dancing; Injury;Sports; Stress, Psychological
Keywords: Dancing; Injury; Qualitative research; Injury, sports; Dancer; Anxiety; Fear; Prevention; Quality Assurance, Health Care; Stress, Psychological; Ballet; Modern dancing
MeSH Terms: conditions — Wounds and Injuries; Athletic Injuries; Stress, Psychological; Anxiety Disorders | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dancers: Dancers or dance students who pracitce at least 8 hours/week
  Interventions: Other: Focus group or interview

INTERVENTIONS:
Other: Focus group or interview — Focus groups and qualitative interview will be conducted with dancers investigating thoughts, beliefs and behaviors related to injury. Individual interviews (in presence or online) will be hold as alternative if it will not be possible (due to logistical or personal problems) to participate in a focus group or if the number of people who would have agreed to participate in that focus group is less than 3

SUMMARY:
This qualitative, cross-sectional study aims at describing the experience of Italian dancers with injury.

Dancers face a high risk of sustaining one or more injuries during their career (87-94%), which may lead to physical, psychological, and socioeconomic consequences affecting dancer's lives and careers both short and long-term.

Dancers report fearing injury and its consequences and believing in the existence of a stigma around injury and injured colleagues; many of them also try to self-manage pain and delay reporting injuries to healthcare professionals, possibly making its outcomes worse.

This study will collect data from dancers via focus groups and individual interviews, investigating dancers' experiences, thoughts, and beliefs about injury. Records from the interviews will be transcribed ad verbatim and analyzed using the framework method to synthetize the data and highlight the most meaningful content.

Understanding dancers' thoughts and behaviors regarding past or possible future injuries may be beneficial in improving treatment efficacy and designing adequate education and prevention strategies. It may also help raise awareness of dancers' complex and unique needs, and the importance of having accessible, specialized professionals around dance companies and schools.

DETAILED DESCRIPTION:
The dance world is a complex setting characterized by high injury risk, high competitivity, high prevalence of risk-taking behaviors, low socio-economic support and a cultural exaltation of sacrifice and pushing through pain and injury to go dancing. With the rapid development of dance medicine and science in the last few decades, it has been highlithed that dancers face a high risk of sustaining one or more injuries during their career, which often come with harsh physical, psychological and economic consequences.

Recent studies show that a great number of dancers are afraid of injury and believe in the existence of a "stigma" surrounding injury and injured colleagues; those who stop dancing report feelings of isolation, insecurity and low confidence in full recovery.

In addition to this, dancers often delay seeking medical attention and treatment when they suspect an injury and try to keep dancing through pain (ignoring symptoms, modifying their activity and/or using painkillers) or relay on non-medical specialist, possibly worsening the outcomes of said injury.

There seems to be a negative halo surrounding injury, and also a mismatch between the high medical needs of the dance population and their healthcare-seeking behaviors.

Research shows trends are slowly getting better in context where dance medicine is well developed and easily available to dancers, especially in larger dance companies, but there is still much to be done.

This research aims to describe the experience of dancers with injury to understand the reasons behind their thoughts and behaviors. Untangling the complex dancer-injury-context relationship will help in in improving care delivery efficacy and designing adequate and specific education and prevention strategies.

Collecting data from questionaires and semi-structured interviews, this study will investigate:

* What is perceived as "injury" by dancers and what will mean for them to sustain an injury
* How dancers cope with pain and behave when suspecting an injury
* What dancers think of a colleague who has to stop dancing because of an injury, and what role their specific context (teachers, choreographers, caregivers) play in this
* What dancers think will help in reducing injury risk and bargain, if they believe it possible
* The functional status of dancers taking part in the interview, past or present history of injury, Dance Functional Outcome Score (DFOS) This research will employ qualitative methods to collect and analyze data, allowing in-depht exploration of dancers' opinions and experiences.

Volounteer participants will be recruited from dance schools and companies in different locations around Italy.

Focus group interviews will be arranged within small groups of dancers (4-8 at a time), accommodating participants in individual interviews if logistical or personal challenges arise. Anagraphic data and the DFOS will be collected by questionnaires prior to the interviews.

The interviews will be sistematically recorded and transcribed ad verbatim to undergo the process of qualitative analysis using the framework method, allowing to extract the most recurrent themes and highlight meaningful insights.

Results from this research may help in improving care delivery efficacy and designing adequate and specific education and prevention strategies, promoting dancers' physical and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who train in dance (any style) 8 hours/week or more
* Individuals who ususally train in dance 8 hours/week or more but have temporarilly suspended their activity due to injury or other condition

Exclusion Criteria:

* Individuals who do not wish to partecipate or do not give consent to data treatment
* Individuals who do not speak Italian or English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dancers and pre-professional dance students who train 8 hours/week or more
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Experience and perception of injury amongst dancers | 120 minutes
  Evaluation of dancers' experience and perception of injury, including the meaning of the term "injury", description of injury-related behaviors that happend in the past or may be applied in the future, description of injury-related emotions (such as fear), and thoughts.
  Information will be collected via semi-structured interviews and then undergo qualitative analisys

SECONDARY OUTCOMES:
Understanding of injury prevention and pain management amongst dancers | 120 minutes
  Evaluation of what dancers believe to be injury prevention and how they manage pain in their activity. Information will be collected via semi-structured interviews and then undergo qualitative analisys

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Bigi, BA, Principal Investigator — University of Siena

IPD SHARING:
Plan to Share IPD: Undecided
Recording will be anonymised and transcripted verbatim. This anonimised material could be shared with other researchers on request

REFERENCES:
- [Background] McEwen K, Young K. Ballet and pain: reflections on a risk-dance culture. Qualitative Research in Sport, Exercise and Health (2011) 3:2, 152-173
- [Result] Vassallo AJ, Pappas E, Stamatakis E, Hiller CE. Injury Fear, Stigma, and Reporting in Professional Dancers. Saf Health Work. 2019 Sep;10(3):260-264. doi: 10.1016/j.shaw.2019.03.001. Epub 2019 Mar 23. PMID 31497323
- [Result] Air M. Health care seeking behavior and perceptions of the medical profession among pre- and post-retirement age Dutch dancers. J Dance Med Sci. 2009;13(2):42-50. PMID 19508808